CLINICAL TRIAL: NCT01397266
Title: Effect of Magnetic Stimulation Repetitive Transcranial on Impulsivity in Cocaine Dependence.
Brief Title: Study of the Effect of Magnetic Stimulation Repetitive Transcranial on Impulsivity in Cocaine Dependence
Acronym: TMSCOCAINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Study of the Effect of Magnetic Stimulation Repetitive Transcranial on Impulsivity in Cocaine Dependence, USaoPauloGH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1339/09
Record Dates: First submitted 2011-05-13; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2010-08

CONDITIONS: Cocaine Dependence
Keywords: Transcranial Magnetic Stimulation; Cocaine; impulsivity; rating scale
MeSH Terms: conditions — Cocaine-Related Disorders; Impulsive Behavior | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active TMS (Active Comparator): active rTMS delivered to the left dorsolateral prefrontal cortex
  Interventions: Procedure: Transcranial Magnetic Stimulation
- Placebo TMS (Placebo Comparator): PLACEBO rTMS delivered to the left dorsolateral prefrontal cortex
  Interventions: Procedure: Placebo TMS

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — ACTIVE rTMS delivered to the left dorsolateral prefrontal cortex
  Other Names: TMS
  Arms: Active TMS
Procedure: Placebo TMS — PLACEBO rTMS delivered to the left dorsolateral prefrontal cortex
  Other Names: TMS
  Arms: Placebo TMS

SUMMARY:
In a randomized, double-blind controlled trial the investigators will evaluate the efficacy of rTMS in reducing impulsivity for cocaine addicts through - Quantitative and qualitative analysis - such behavior and possible behavioral consequences related.

DETAILED DESCRIPTION:
reduction of the rating impulsivity

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of the cocaine dependence syndrome, alone or in combination with abuse of alcohol and nicotine dependence (DSM IV, 1994; SCID-P, 1994).
2. 20 days or less withdrawal
3. 18-35 years old.
4. If female, to be using contraception (barrier, oral contraceptive, IUD, surgical sterilization).
5. Fixed residential address in Sao Paulo

Exclusion criteria:

1. Other Mental Disorders (DSM IV, 1994; SCID-P, 1994).
2. organic brain disease, neurosurgery to implant metal clip or epilepsy.
3. severe uncontrolled clinical comorbidity.
4. use current or within last six months of psychotropic drugs in general, except for Clonazepam dose of up to four mg / day.
5. Changes clinically significant laboratory findings. 13
6. Condition or situation to which in the opinion of the investigator put the patient at risk significant, which may confound the results, or interfere substantially in individual's participation in the study.
7. Mandate that mandating the judicial treatment for cocaine dependence

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-01 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The Short PROMIS Questionnaire | 2 months
  The SPQ is a 160-question paper that counsellors and researchers can use to measure an individual's level of addictive tendency in each of sixteen distinct behavioural areas. Will be applied at the following times:
  T0 (weeks 0 - immediately prior to the rTMS) T1 (4 weeks, after four weeks of treatment with rTMS) and T2 (8 weeks, four weeks after completing treatment).
  The improvement rate of 10% or more, will be our primary measure of efficacy. T0 (

CONTACTS AND LOCATIONS:
Overall Officials: Adan Jardim, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Department and Institute of Psychiatry, General Hospital, University of São Paulo Medical School, São Paulo, São Paulo, Brazil